CLINICAL TRIAL: NCT02318277
Title: A Phase 1/2 Study Exploring the Safety, Tolerability, and Efficacy of Epacadostat (INCB024360) in Combination With Durvalumab (MEDI4736) in Subjects With Selected Advanced Solid Tumors (ECHO-203)
Brief Title: A Study of Epacadostat (INCB024360) in Combination With Durvalumab (MEDI4736) in Subjects With Selected Advanced Solid Tumors (ECHO-203)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 24360-203 / ECHO-203
Record Dates: First submitted 2014-11-19; First posted 2014-12-17 (Estimated); Results first posted 2020-12-29 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Solid Tumors; Head and Neck Cancer; Lung Cancer; UC (Urothelial Cancer)
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms | interventions — durvalumab; epacadostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MEDI4736 + INCB024360 (Experimental): MEDI4736 at selected dose levels every 2 weeks + INCB024360 25 mg BID as starting dose, followed by dose escalations until MTD or PAD is identified
  Interventions: Drug: MEDI4736; Drug: INCB024360

INTERVENTIONS:
Drug: MEDI4736 — MEDI4736 administered intravenously (IV) every two weeks (q2w)
Drug: INCB024360 — INCB024360: Oral daily dosing

SUMMARY:
The purpose of this study is to explore the safety, tolerability, pharmacokinetics, immunogenicity and preliminary efficacy of INCB024360 administered in combination with MEDI4736 in subjects with selected advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, age 18 years or older
* Histologically or cytologically confirmed diagnosis of selected locally advanced or metastatic solid tumors
* Must have failed at least 1 prior treatment regimen for locally advanced or metastatic disease or be intolerant to treatment or refuse standard treatment

Exclusion Criteria:

* Laboratory and medical history parameters not within protocol-defined range
* Participation in any other study in which receipt of an investigational study drug occurred within 28 days or 5 half-lives (whichever is longer) prior to first dose
* Prior treatment with immune checkpoint inhibitors (eg, anti-CTLA-4, anti-PD-1, anti-PD-L1, and any other antibody or drug specifically targeting T-cell co-stimulation) or an IDO inhibitor (exception is tumor types in which a PD-1 pathway targeted agent is approved, e.g. melanoma, non-small cell lung cancer.)
* Receipt of any anticancer medication in the 21 days prior to receiving the first dose of study medication
* Has an active or inactive autoimmune process
* Evidence of interstitial lung disease or active, non-infectious pneumonitis
* Prior radiotherapy within 2 weeks of initiating treatment; Must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis
* Untreated central nervous system (CNS) metastases or CNS metastases that have progressed
* Currently pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2020-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lance Leopold, MD, Study Director — Incyte Corporation
Locations (13):
- United States (13):
  - San Francisco, California
  - Denver, Colorado
  - Miami, Florida
  - Port Saint Lucie, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Louisville, Kentucky
  - Durham, North Carolina
  - Huntersville, North Carolina
  - Winston-Salem, North Carolina
  - Dallas, Texas
  - Houston, Texas

REFERENCES:
- [Derived] Naing A, Algazi AP, Falchook GS, Creelan BC, Powderly J, Rosen S, Barve M, Mettu NB, Triozzi PL, Hamm J, Zhou G, Walker C, Dong Z, Patel MR. Phase 1/2 study of epacadostat in combination with durvalumab in patients with metastatic solid tumors. Cancer. 2023 Jan 1;129(1):71-81. doi: 10.1002/cncr.34512. Epub 2022 Oct 30. PMID 36309837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 13 study sites in the United States. Participants were enrolled at 12 study sites.
Pre-assignment Details: A total of 235 participants were screened and 59 participants were screen failures. A total of 176 participants ( 34 participants in Phase 1 and 142 in Phase 2) were enrolled in the study. Study enrollment was permanently discontinued on 24 Apr 2018 as a strategic decision. At the time of data cut-off, 28 Aug 2019, 1 participant was ongoing.
Groups:
- Phase I : Epacadostat (25 mg) + Durvalumab (3 mg/kg): Epacadostat (25 mg) oral twice-daily (BID) dosing in combination with durvalumab (3 mg/kg) administered intravenously (IV) on Day 1 of each 14 day cycle.
- Phase I : Epacadostat (25 mg) + Durvalumab (10 mg/kg): Epacadostat (25 mg) oral twice-daily (BID) dosing in combination with durvalumab (10 mg/kg) administered intravenously (IV) on Day 1 of each 14 day cycle.
- Phase I : Epacadostat (50 mg) + Durvalumab (10 mg/kg): Epacadostat (50 mg) oral twice-daily (BID) dosing in combination with durvalumab (10 mg/kg) administered intravenously (IV) on Day 1 of each 14 day cycle.
- Phase I : Epacadostat (75 mg) + Durvalumab (10 mg/kg): Epacadostat (75 mg) oral twice-daily (BID) dosing in combination with durvalumab (10 mg/kg) administered intravenously (IV) on Day 1 of each 14 day cycle.
- Phase I : Epacadostat (100 mg) + Durvalumab (10 mg/kg): Epacadostat (100 mg) oral twice-daily (BID) dosing in combination with durvalumab (10 mg/kg) administered intravenously (IV) on Day 1 of each 14 day cycle.
- Phase I : Epacadostat (300 mg) + Durvalumab (10 mg/kg): Epacadostat (300 mg) oral twice-daily (BID) dosing in combination with durvalumab (10 mg/kg) administered intravenously (IV) on Day 1 of each 14 day cycle.
- Phase II : Epacadostat (100 mg) + Durvalumab (10 mg/kg): Epacadostat (100 mg) oral twice-daily (BID) dosing in combination with durvalumab (10 mg/kg) administered intravenously (IV) on Day 1 of each 14 day cycle in select tumor types.
- Phase II : Epacadostat (300 mg) + Durvalumab (10 mg/kg): Epacadostat (300 mg) oral twice-daily (BID) dosing in combination with durvalumab (10 mg/kg) administered intravenously (IV) on Day 1 of each 14 day cycle in select tumor types.
Period: Overall Study
Arm/Group | Phase I : Epacadostat (25 mg) + Durvalumab (3 mg/kg) | Phase I : Epacadostat (25 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (50 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (75 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (300 mg) + Durvalumab (10 mg/kg) | Phase II : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase II : Epacadostat (300 mg) + Durvalumab (10 mg/kg)
Started | 6 | 3 | 4 | 4 | 8 | 9 | 49 | 93
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 3 | 4 | 4 | 8 | 9 | 49 | 93
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 1 | 6 | 14
Not completed — Participant trial terminated by sponsor | 0 | 0 | 1 | 0 | 1 | 2 | 5 | 16
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 4
Not completed — Death | 5 | 3 | 1 | 4 | 6 | 5 | 34 | 58
Not completed — Transitioned to Hospice | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population who are enrolled in Phase 1 and 2 part of the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I : Epacadostat (25 mg) + Durvalumab (3 mg/kg) | Phase I : Epacadostat (25 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (50 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (75 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (300 mg) + Durvalumab (10 mg/kg) | Phase II : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase II : Epacadostat (300 mg) + Durvalumab (10 mg/kg) | Total
Number analyzed (Participants) | 6 | 3 | 4 | 4 | 8 | 9 | 49 | 93 | 176
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.8 (4.79) | 75.7 (7.23) | 65.3 (9.07) | 72.3 (7.59) | 58.6 (8.65) | 63.4 (7.75) | 60.2 (13.24) | 64 (10.27) | 63.3 (11.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 1 | 1 | 5 | 19 | 25 | 57
  Male | 3 | 1 | 3 | 3 | 7 | 4 | 30 | 68 | 119
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 3 | 4 | 4 | 7 | 9 | 41 | 83 | 157
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 5 | 11
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 4
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 7
  Not Hispanic or Latino | 4 | 3 | 4 | 3 | 8 | 9 | 46 | 87 | 164
  Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 : Number of Treatment-Emergent Adverse Events (TEAE)
Description: Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment
Time Frame: Duration of study treatment and up to 90 days after the last dose [approximately 3 years]
Population: The Phase 1 safety population includes all subjects enrolled in the Phase 1 portion of the study who received at least 1 dose of INCB024360 or MEDI4736. Treatment groups were determined according to the actual treatment the subject received on Day 1 regardless of the actual study drug the subject received during participation in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I : Epacadostat (25 mg) + Durvalumab (3 mg/kg) | Phase I : Epacadostat (25 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (50 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (75 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (300 mg) + Durvalumab (10 mg/kg)
Number analyzed (Participants) | 6 | 3 | 4 | 4 | 8 | 9
Participants | 6 | 3 | 4 | 4 | 8 | 9

2. Primary Outcome: Phase 2: Objective Response Rate (ORR) as Determined by Radiographic Disease Assessments Per Modified Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: ORR was defined as the percentage of participants having a complete response (CR) or partial response (PR) as determined by investigator assessment of radiographic disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Time Frame: Measured every 8 weeks for duration of study treatment [approximately 12 months]
Population: Intent-to-Treat Population : All subjects who are enrolled in the Phase 2 portion of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase II : Epacadostat (300 mg) + Durvalumab (10 mg/kg)
Number analyzed (Participants) | 49 | 93
Participants | 6 | 12

3. Secondary Outcome: Phase 1: Objective Response Rate (ORR) as Determined by Radiographic Disease Assessments Per Modified RECIST v1.1
Description: as for outcome 2
Time Frame: Measured every 8 weeks for duration of study treatment [approximately 6 months]
Population: Intent-to-Treat Population: All subjects who are enrolled in the Phase 1 portion of the study. Treatment groups for this population were defined according to the treatment assignment at the time of enrollment on Day 1 regardless of the actual study drug the subject received during his/her continued participation in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I : Epacadostat (25 mg) + Durvalumab (3 mg/kg) | Phase I : Epacadostat (25 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (50 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (75 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (300 mg) + Durvalumab (10 mg/kg)
Number analyzed (Participants) | 6 | 3 | 4 | 4 | 8 | 9
Participants | 1 | 0 | 1 | 0 | 1 | 2

4. Secondary Outcome: Phase 2: Number of Treatment-Emergent Adverse Events
Description: as for outcome 1
Time Frame: Continuously for duration of study treatment and up to 90 days after the last dose [approximately 3 years]
Population: The Phase 2 safety population includes all subjects enrolled in the Phase 2 portion of the study who received at least 1 dose of INCB024360 or MEDI4736.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase II : Epacadostat (300 mg) + Durvalumab (10 mg/kg)
Number analyzed (Participants) | 49 | 93
Participants | 49 | 93

5. Secondary Outcome: Phase 1 and 2: Durability of Response as Measured by the Time From the Earliest Date of Disease Response Until Earliest Date of Disease Progression
Description: Defined as the time from earliest date of disease response until the earliest date of disease progression per RECIST v1.1, or death due to any cause, if occurring sooner than progression.
Time Frame: Measured every 8 weeks for duration of active study treatment [approximately 24 months]
Population: Intent-to-Treat Population: All subjects who are enrolled in the Phase 1 & 2 portion of the study. Treatment groups were defined at the time of enrollment on Day 1 according to the treatment assignment for Phase 1 and according to the tumor type for phase 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I : Epacadostat (25 mg) + Durvalumab (3 mg/kg) | Phase I : Epacadostat (25 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (50 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (75 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (300 mg) + Durvalumab (10 mg/kg) | Phase II : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase II : Epacadostat (300 mg) + Durvalumab (10 mg/kg)
Number analyzed (Participants) | 1 | 0 | 1 | 0 | 1 | 2 | 6 | 12
months | 1.9 [NA to NA] — Upper and Lower bound not estimable due to sample size |  | NA [NA to NA] — Median not estimable due to censoring |  | NA [NA to NA] — Median not estimable due to censoring | NA [25.6 to NA] — Median not estimable due to censoring | 13.8 [8.5 to NA] — Due to the definition of confidence interval in SAS proc lifetest, the time point satisfying the upper bound from the formula happens to be censored, therefore it is not NE | NA [1.9 to NA] — Median duration and Upper bound is not estimable due to due to the many censored observations

6. Secondary Outcome: Phase 1 and 2: Progression-free Survival as Measured by the Duration From the Date of Enrollment Until the Earliest Date of Disease Progression or Death
Time Frame: Measured every 8 weeks for duration of active study treatment [approximately 24 months]
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase I : Epacadostat (25 mg) + Durvalumab (3 mg/kg) | Phase I : Epacadostat (25 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (50 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (75 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (300 mg) + Durvalumab (10 mg/kg) | Phase II : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase II : Epacadostat (300 mg) + Durvalumab (10 mg/kg)
Number analyzed (Participants) | 6 | 3 | 4 | 4 | 8 | 9 | 49 | 93
Months | 2.4 [1.3 to 7.3] | 12.0 [1.8 to NA] — Due to the definition of confidence interval in SAS proc lifetest, the time point satisfying the upper bound from the formula happens to be censored, therefore it is not estimable | 1.9 [1.1 to NA] — Due to the definition of confidence interval in SAS proc lifetest, the time point satisfying the upper bound from the formula happens to be censored, therefore it is not estimable | 1.7 [0.5 to 5.9] | 4.1 [0.7 to NA] — Due to the definition of confidence interval in SAS proc lifetest, the time point satisfying the upper bound from the formula happens to be censored, therefore it is not estimable | 2.5 [1.1 to 27.2] | 1.9 [1.7 to 2.3] | 2.1 [1.9 to 3.7]

7. Secondary Outcome: Phase 1 and 2: Pharmacokinetics (PK) of INCB024360 as Measured by Peak Concentration
Time Frame: Pre dose, 0.5, 1,2, 4.6.& 8 hrs Post dose on C1D1,C1D8,C2D1
Population: The PK evaluable population will include all subjects who received at least 1 dose of INCB024360 and provided at least 1 post dose plasma sample (1 PK/PD measurement). Phase I : Epacadostat (25 mg) + Durvalumab (3 mg/kg)" Arm/Group were combined with the data collected from participants in the "Phase I : Epacadostat (25 mg) + Durvalumab (10 mg/kg)" Arm/Group for PK Analysis.
Measure: Mean (Standard Deviation); unit: nM
Groups:
- Phase I : Epacadostat (25 mg) + Durvalumab: Epacadostat (25 mg) oral twice-daily (BID) dosing in combination with durvalumab (3 or 10 mg/kg) administered intravenously (IV) on Day 1 of each 14 day cycle.
Arm/Group | Phase I : Epacadostat (25 mg) + Durvalumab | Phase I : Epacadostat (50 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (75 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (300 mg) + Durvalumab (10 mg/kg) | Phase II : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase II : Epacadostat (300 mg) + Durvalumab (10 mg/kg)
Number analyzed (Participants) | 8 | 3 | 3 | 7 | 7 | 38 | 36
nM | 273 (65.3) | 248 (135) | 604 (493) | 727 (403) | 2660 (1200) | 960 (499) | 2500 (1190)

8. Secondary Outcome: Phase 1 and 2: Pharmacokinetics (PK) of INCB024360 as Measured by Time to Maximal Observed Concentration
Time Frame: Pre dose, 0.5, 1,2, 4.6.& 8 hrs Post dose on C1D1,C1D8,C2D1
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Phase I : Epacadostat (25 mg) + Durvalumab | Phase I : Epacadostat (50 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (75 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (300 mg) + Durvalumab (10 mg/kg) | Phase II : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase II : Epacadostat (300 mg) + Durvalumab (10 mg/kg)
Number analyzed (Participants) | 8 | 3 | 3 | 7 | 7 | 38 | 36
hours | 2.0 [1.0 to 2.2] | 2.0 [1.0 to 3.8] | 1.9 [0.017 to 3.9] | 2.0 [0.92 to 6.0] | 3.3 [1.2 to 6.0] | 2.0 [0.0 to 5.7] | 2.1 [0.52 to 5.5]

9. Secondary Outcome: Phase 1 and 2: Pharmacokinetics (PK) of INCB024360 as Area Under the Concentration-time Curve
Time Frame: Pre dose, 0.5, 1,2, 4.6.& 8 hrs Post dose on C1D1,C1D8,C2D1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: h*nM
Arm/Group | Phase I : Epacadostat (25 mg) + Durvalumab | Phase I : Epacadostat (50 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (75 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (300 mg) + Durvalumab (10 mg/kg) | Phase II : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase II : Epacadostat (300 mg) + Durvalumab (10 mg/kg)
Number analyzed (Participants) | 8 | 3 | 3 | 7 | 7 | 36 | 34
h*nM | 1040 (345) | 1580 (739) | 3090 (1880) | 3650 (2710) | 15400 (6770) | 4130 (1960) | 12200 (5950)

10. Secondary Outcome: Phase 1 and 2: Immunogenicity of MEDI4736 as Measured by the Number and Percentage of Subjects Who Develop Detectable Anti-drug Antibodies (ADAs)
Time Frame: Measured at defined study visits from Cycle 1 Day 1 through cycle 2 [approximately 2 weeks].
Population: Evaluable Patients Post-Baseline: Treatment-Induced ADA - Patients who had baseline negative ADA result who developed anti-drug antibodies at any time after initial drug administration.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I : Epacadostat (75 mg) + Durvalumab (10 mg/kg)Edit: Epacadostat (75 mg) oral twice-daily (BID) dosing in combination with durvalumab (10 mg/kg) administered intravenously (IV) on Day 1 of each 14 day cycle.
- Phase I : Epacadostat (300 mg) + Durvalumab (10 mg/kg)Edit: Epacadostat (300 mg) oral twice-daily (BID) dosing in combination with durvalumab (10 mg/kg) administered intravenously (IV) on Day 1 of each 14 day cycle.
- Phase 2 Stage 1: Epacadostat (100 mg) + Durvalumab (10 mg/kg): Epacadostat (100 mg) oral twice-daily (BID) dosing in combination with durvalumab (10 mg/kg) administered intravenously (IV) on Day 1 of each 14 day cycle to determine maximum Tolerated dose (MTD) or pharmacologically active dose (PAD).
- Phase 2 Stage 2: Epacadostat (300 mg) + Durvalumab (10 mg/kg): Epacadostat (300 mg) oral twice-daily (BID) dosing in combination with durvalumab (10 mg/kg) administered intravenously (IV) on Day 1 of each 14 day cycle to determine maximum Tolerated dose (MTD) or pharmacologically active dose (PAD).
Arm/Group | Phase I : Epacadostat (25 mg) + Durvalumab (3 mg/kg) | Phase I : Epacadostat (25 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (50 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (75 mg) + Durvalumab (10 mg/kg)Edit | Phase I : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (300 mg) + Durvalumab (10 mg/kg)Edit | Phase 2 Stage 1: Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase 2 Stage 2: Epacadostat (300 mg) + Durvalumab (10 mg/kg)
Number analyzed (Participants) | 4 | 2 | 3 | 3 | 7 | 8 | 36 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Duration of study treatment and up to 90 days after the last dose [approximately 3 years]
Arm/Group | Phase I : Epacadostat (25 mg) + Durvalumab (3 mg/kg) | Phase I : Epacadostat (25 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (50 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (75 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase I : Epacadostat (300 mg) + Durvalumab (10 mg/kg) | Phase II : Epacadostat (100 mg) + Durvalumab (10 mg/kg) | Phase II : Epacadostat (300 mg) + Durvalumab (10 mg/kg)
All-Cause Mortality (participants affected / at risk) | 5/6 | 3/3 | 1/4 | 4/4 | 6/8 | 5/9 | 35/49 | 58/93
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/3 | 2/4 | 0/4 | 4/8 | 3/9 | 20/49 | 54/93
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 4/4 | 4/4 | 8/8 | 9/9 | 48/49 | 87/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I : Epacadostat (25 mg) + Durvalumab (3 mg/kg) (N=6) | Phase I : Epacadostat (25 mg) + Durvalumab (10 mg/kg) (N=3) | Phase I : Epacadostat (50 mg) + Durvalumab (10 mg/kg) (N=4) | Phase I : Epacadostat (75 mg) + Durvalumab (10 mg/kg) (N=4) | Phase I : Epacadostat (100 mg) + Durvalumab (10 mg/kg) (N=8) | Phase I : Epacadostat (300 mg) + Durvalumab (10 mg/kg) (N=9) | Phase II : Epacadostat (100 mg) + Durvalumab (10 mg/kg) (N=49) | Phase II : Epacadostat (300 mg) + Durvalumab (10 mg/kg) (N=93)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angiopathy (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Contrast media reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (7) | 4 (4)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 3 (3)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I : Epacadostat (25 mg) + Durvalumab (3 mg/kg) (N=6) | Phase I : Epacadostat (25 mg) + Durvalumab (10 mg/kg) (N=3) | Phase I : Epacadostat (50 mg) + Durvalumab (10 mg/kg) (N=4) | Phase I : Epacadostat (75 mg) + Durvalumab (10 mg/kg) (N=4) | Phase I : Epacadostat (100 mg) + Durvalumab (10 mg/kg) (N=8) | Phase I : Epacadostat (300 mg) + Durvalumab (10 mg/kg) (N=9) | Phase II : Epacadostat (100 mg) + Durvalumab (10 mg/kg) (N=49) | Phase II : Epacadostat (300 mg) + Durvalumab (10 mg/kg) (N=93)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 5 (5) | 10 (10)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 10 (13)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 6 (11)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 11 (11) | 11 (13)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 6 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 6 (7) | 9 (15)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (5) | 11 (13)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 7 (7) | 10 (10)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 12 (13)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 15 (18)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Blood prolactin abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Blood testosterone decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Catheter site discharge (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 6 (7) | 8 (10)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 11 (11) | 20 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 7 (9) | 19 (26)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 9 (12) | 26 (26)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 14 (17)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (4) | 10 (15) | 22 (28)
Dizziness (Nervous system disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 9 (10)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (6)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (7) | 13 (18)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 7 (9)
Fatigue (General disorders) | 4 (4) | 1 (1) | 2 (3) | 2 (2) | 3 (5) | 2 (2) | 25 (28) | 50 (54)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Foreign body aspiration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (3)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 6 (8) | 16 (20)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 7 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 5 (12) | 8 (23)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (6)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 6 (8)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 5 (6)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (5) | 6 (6)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypogonadism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 8 (8)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 4 (4) | 8 (10)
Hypotension (Vascular disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 7 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 16 (16)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 9 (10)
Lower urinary tract symptoms (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (5)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 5 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 14 (16)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 4 (6) | 3 (4) | 13 (19) | 28 (33)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 7 (7) | 5 (5)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (5)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 5 (5) | 9 (10)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 8 (8)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (4) | 4 (5) | 13 (17)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (2) | 11 (12) | 10 (15)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 10 (11)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 1 (2) | 9 (14) | 10 (13)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Serotonin syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 8 (9)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 3 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 9 (9)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (9)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 5 (6)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (5) | 7 (10) | 17 (20)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 6 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT02318277/Prot_000.pdf
  • Statistical Analysis Plan (2014-11-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT02318277/SAP_001.pdf